CLINICAL TRIAL: NCT06004037
Title: A Phase 2a, Open-label, Single-arm, Multi-center Study to Evaluate the Efficacy and Safety of LCB01-0371 (Delpazolid) as Add-on Therapy in Patients With Refractory Mycobacterium Abscessus Complex Pulmonary Disease
Brief Title: Study to Evaluate the Efficacy of Delpazolid as Add-on Therapy in Refractory Mycobacterium Abscessus Complex
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCB01-0371-2004
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Nontuberculous Mycobacterium Infection; Mycobacterium Abscessus Infection
Keywords: NTM; MABC; MABC-PD; rapid growers
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — delpazolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- delpazolid (Experimental): In addition to background therapy for MABC, patients will be given orally three tablets (400 mg/tablet) of LCB01-0371 for 12 weeks.
  Interventions: Drug: Delpazolid

INTERVENTIONS:
Drug: Delpazolid — Three tablets (400 mg/tablet) of delpazolid will be orally administered once daily for 12 weeks.
  After 3 months (12 weeks) of administration, if the investigator determines that there are clinical benefits, an additional extended treatment of up to 9 months (40 weeks) may be given, amounting to 1 year of treatment in total.
  Other Names: LCB01-0371

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of delpazolid add-on therapy in Patients with Refractory Mycobacterium abscessus Complex Pulmonary disease

DETAILED DESCRIPTION:
Delpazolid, which demonstrates effects similar to other oxazolidinone-class drugs and has confirmed good safety, aims to evaluate its efficacy in MABC-PD patients who are unresponsive to guideline-based treatments

ELIGIBILITY:
Inclusion Criteria:

* Pre-screening: Adults aged 19 years or above
* Pre-screening: Patients diagnosed with MABC (including subspecies abscessus, bolletii, and massiliense) pulmonary disease in radiologic and microbiologic evaluations
* LCB01-0371 MIC ≤ 8 μg/mL for MABC
* Patients who continue to show positivity for MABC even after treatments based on the guidelines of ATS/ERS/ESCMID/IDSA for at least 6 months prior to screening, and who meet all of the following criteria:

  1. Patients who have been confirmed positive at least once in the last sputum or bronchoscopy sample culture performed prior to screening
  2. Patients who have not achieved culture conversion (at least 3 consecutive negative mycobacteria cultures in the sputum or bronchoscopy sample collected at an interval of at least 4 weeks) within 6 months prior to screening
* Patients who can voluntarily expectorate sputum at screening
* Patients with a life expectancy of 12 weeks or more
* Patients with adequate organ function who meet the following criteria:

  1. Hemoglobin > 9.0 g/dL (without transfusion within 2 weeks prior to measurement)
  2. Absolute neutrophil count ≥ 1,500/µL (without administration of G-CSF within 2 weeks prior to measurement)
  3. Platelet ≥ 100,000/µL
  4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
  5. Alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 2.5 × ULN
  6. Serum creatinine ≤ 1.5 × ULN or creatinine clearance >30 mL/min (calculated with the Cockcroft-Gault formula)
* Patients who voluntarily provided a written consent to participate in the clinical study

Exclusion Criteria:

* Patients who cannot swallow the study drug tablet due to dysphagia, nasogastric tube insertion, etc.
* Patients diagnosed with cystic fibrosis
* Patients who have received a lung transplant
* Patients with disseminated or extrapulmonary nontuberculous mycobacteria
* Patients with known active pulmonary tuberculosis
* Patients with NTM infections other than MABC
* Patients with an active pulmonary malignancy within 1 year prior to screening or Patients with other malignancies that require chemotherapy or radiotherapy
* Patients who has received linezolid for MABC treatment within 3 months prior to screening
* Patients with known HIV positivity or a suspected infection thereof or Patients with a known active hepatitis B or C infection
* Patients who currently have a clinically significant cardiovascular disease

  1. Patients with severe cardiac failure (New York Heart Association [NYHA] class III/IV) that occurred within 24 weeks prior to screening
  2. Patients with pulmonary embolism or deep venous thrombosis that occurred within 24 weeks prior to screening
* Patients whose multidrug therapy for treatment of MABC was changed within 4 weeks prior to screening (Discontinuation, dose adjustment, change of administration route, etc., are allowed.)
* Patients for whom the administration of contraindicated concomitant drugs that correspond to the following cannot be discontinued during the clinical study or for whom their administration is necessary

  1. Administration of a new antibacterial agent for the prioritized treatment of NTM, especially MABC, other than background therapy
  2. Monoamine oxidase inhibitors
  3. Serotonin reuptake inhibitor or serotonin 5-HT1 receptor agonists
  4. Meperidine or buspirone
  5. Drugs that lower epilepsy threshold; tramadol, etc.
  6. Tricyclic Antidepressant
  7. Other investigational products: If there is a history of administration within 30 days prior to screening, it falls under the exclusion criteria.
* Pregnant or breastfeeding women and women of childbearing potential who do not agree to practice appropriate contraceptive methods*:

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
semi-quantitative scale (SQS) change versus baseline | 12 weeks
  The SQS using liquid media and solid media will be scored a point of 1-7, with lower scores representing a reducing bacterial load.

SECONDARY OUTCOMES:
Change from baseline in SQS | 4 weeks and 8 weeks
  The SQS using liquid media and solid media will be scored a point of 1-7, with lower scores representing a reducing bacterial load.
Sputum culture conversion rate | 12 weeks
  neg culture x3( sputum conversion)
Time to culture conversion | 12 weeks
  from the date of assignment to the first negative result.
Time to positivity in the liquid culture automated system (MGIT) | 12 weeks
  time to detection of positive in MGIT system
Negative sputum culture rate at each time point after baseline | 12 weeks
  negative culture results in MGIT and solid media
Change from baseline in the inflammatory marker | 12 weeks
  erythrocyte sedimentation rate [ESR]) at each time point
Change from baseline in the CT score | 12 weeks
  The CT scan score will be transformed onto a scale of 0-42, with lower scores representing improved lung presentations.
  Descriptive statistics for each point in time are presented, and intra-group comparison of CT score changes at 12 weeks compared to baseline
Quality of Life Questionnaire-Bronchiectasis | 12 weeks
  The QOL-B respiratory symptoms score was transformed onto a scale of 0-100, with higher scores representing a better quality of life.
Six-minute walk test | 12 weeks
  Six-minute walk test
Extended administration | After 12 weeks
  1) SQS at each time point compared to baseline in subjects receiving extended administration
  * The SQS using liquid media and solid media will be scored a point of 1-7, with lower scores representing a reducing bacterial load 2) Inflammatory markers at each time point compared to baseline in subjects receiving extended administration
  * erythrocyte sedimentation rate 3) CT scores at each time point compared to baseline in subjects receiving extended administration
  * The CT scan score will be transformed onto a scale of 0-42, with lower scores representing improved lung presentations.
    4) QOL-B change at each time point compared to baseline in subjects receiving extended administration
  * The QOL-B respiratory symptoms score was transformed onto a scale of 0-100, with higher scores representing a better quality of life.
    5) sputum culture negative conversion at each time point compared to baseline in subjects receiving extended administration
  * negative culture results in MGIT and solid media

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Asan Medical Center, Seoul
  - Bundang Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No